CLINICAL TRIAL: NCT00568152
Title: Effect of Apple Flavanols on Risk of Cardiovascular Disease
Acronym: FLAVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IFR02-2006; 06/Q101/22
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
Keywords: Apples; Dietary intervention; Procyanidins
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low PA apple puree (Experimental): 230grams of low PA apple puree (Golden Delicious) consumed daily for 14 days.
  Interventions: Dietary Supplement: Low PA apple puree
- High PA apple puree (Experimental): High PA apple puree (Mitchalin) 230grams consumed daily for 14 days
  Interventions: Dietary Supplement: High PA apple puree
- Aspirin (Placebo Comparator): 75mg dispersable aspirin taken daily for 14 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Dietary Supplement: Low PA apple puree — Golden Delicious apple puree 230grams consumed daily for 14 days
  Arms: Low PA apple puree
Dietary Supplement: High PA apple puree — High PA apple puree (Mitchalin) consumed daily for 14 days
  Arms: High PA apple puree
Drug: Aspirin — 75mg dispersable aspirin taken daily for 14 days
  Arms: Aspirin

SUMMARY:
A randomised three period cross over trial will be carried out in adults (19-64 years) to assess the acute and chronic effects of a large dose of apple procyanidin (PA) compared with a low dose of apple PA (negative control) and aspirin (positive control), on platelet function and other risk factors of cardiovascular disease. Platelet function will be assessed prior to a run in diet and at the start and end of each intervention. Volunteers will be assigned at random to consume 230grams of low PA apple puree or high PA apple puree or aspirin (75mg) each day for 2 weeks followed by a minimum 14 day wash out.

Hypothesis: Consuming apple PA reduces platelet function consistent with reduced risk of cardiovascular disease.

DETAILED DESCRIPTION:
A randomised 3-period cross-over trial will be carried out to assess the acute and chronic effects of a large dose of apple PA compared with a low dose of apple PA (negative control) and aspirin (positive control), on platelet function (flow cytometry) and other risk factors of CVD (endothelial function, plasma antioxidants, inflammatory markers, lipid profile). Once recruited, volunteers will be assigned at random to consume 230g of low PA apple puree or high PA apple puree or aspirin (75mg) each day for 14 days in period 1. Following a minimum 14 day wash-out volunteers will then be crossed over for period 2 and after another 14-day wash-out volunteers will be crossed over to complete period 3 of the intervention (flow chart I). The acute effect of each treatment will be investigated on day 15 of each period. A fasting blood sample will be obtained prior to consumption of a standard breakfast and the apple puree or aspirin. Further blood samples will then be obtained at 2, 6 and 24 hours post-dosing. The chronic effect of all three treatments will be determined by measuring CVD risk factors in fasting blood samples obtained on day 1, 15 and 29. Flow chart II provides a more detailed overview of the design of each period which is identical for the apple puree treatments and differs only in the omission of urine collections and PWV measurements for the aspirin period. During the apple puree interventions phenolic acids will be analysed in 24-hour urine pools collected on the day prior to the start of each period, as well as on day 14, 15, and 28. PWV measurements will be carried on day 15 and 29 after a 12-hour overnight fast for each of the 2 apple intervention periods.

For the intervention to be successful it is necessary to exclude some food sources that contribute significantly to total PA intake (e.g. cocoa, berries, grapes, red wine, apples, legumes) and limit other PA food sources (tea/coffee) to levels that support compliance and are unlikely to mask any effects of the intervention. Because of its well documented effect on platelet function alcohol will be restricted to a maximum of 2 units per day and excluded completely for the 48 hours prior to blood sampling appointments. Oily fish consumption will be limited to 2 portions per week and will not be allowed for 48 hours prior to blood sampling. These dietary restrictions may have significant effects on platelet function in individuals that consume these foods regularly. Therefore, dietary restrictions will apply during a 14-day run-in diet prior to and for the duration of each intervention period. Platelet function will be assessed prior to the start of the run-in diet as well as at the start and end of each PA/aspirin intervention (flow chart II).

Male and female volunteers aged 19 to 64 will be recruited and screened for eligibility for up to 2 months prior to the start of the intervention. Those meeting the study criteria will be randomly assigned to one out of the six possible treatment orders, i.e. ABC, ACB, BAC, CAB, BCA, CBA. Randomisation will be stratified by sex.

Volunteers will be given a user friendly booklet (Run-in diet/Apple/Aspirin diary) for each intervention period to record apple puree/aspirin consumption and volunteers will also be prompted to record their alcohol, tea/coffee and oily fish intake (Annex 2). Foods not allowed during each intervention period are listed. Volunteers will be reminded not to consume oily fish (as listed), alcohol, coffee and tea 48 hours prior to a blood sampling appointment.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 19-64

Exclusion Criteria:

* Smokers, very low or high pressure (<90/50 or <95/55 if symptomatic or >160/100), BMI <18.5 or >35, pregnant or have been pregnant in last 12 months, diagnosed with gastrointestinal disease, history of ulcers and gastrointestinal bleeding, diagnosed with a long term illness requiring active treatment, history of stroke, on regularly prescribed medication known to have a profound effect on cardiovascular disease risk factors, using non steroidal anti inflammatory cream, sufferers of asthma or hay fever, known intolerance to aspirin, allergic to apples or birch pollen, regular use of aspirin, antacids or laxatives, unwillingness to discontinue specific dietary or herbal supplements less than 1 month prior to the start of the study, blood donation within 16 weeks of the first study sample, antibiotic use within 4 weeks prior to starting the study, those who receive or plan to receive any type of immunisation within 4 weeks of the start of the study, parallel participation in any other research project.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-05; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The aim of this trial is to investigate the effect of consuming apple PA on platelet function. | 16 weeks

SECONDARY OUTCOMES:
To measure the bioavailability of PA and metabolites from two well characterised apple purees providing a low and high dose of PA. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kroon, Principal Investigator — Quadram Institute Bioscience; Amy Gasper, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institue of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Ambrose JA, Barua RS. The pathophysiology of cigarette smoking and cardiovascular disease: an update. J Am Coll Cardiol. 2004 May 19;43(10):1731-7. doi: 10.1016/j.jacc.2003.12.047. PMID 15145091
- [Background] Donovan JL, Manach C, Rios L, Morand C, Scalbert A, Remesy C. Procyanidins are not bioavailable in rats fed a single meal containing a grapeseed extract or the procyanidin dimer B3. Br J Nutr. 2002 Apr;87(4):299-306. doi: 10.1079/bjnbjn2001517. PMID 12064339
- [Background] DuPont MS, Day AJ, Bennett RN, Mellon FA, Kroon PA. Absorption of kaempferol from endive, a source of kaempferol-3-glucuronide, in humans. Eur J Clin Nutr. 2004 Jun;58(6):947-54. doi: 10.1038/sj.ejcn.1601916. PMID 15164116
- [Background] Gimenez R, Cabrera C, Olalla M, Ruiz MD, Lopez MC. Ascorbic acid in diet supplements: loss in the manufacturing process and storage. Int J Food Sci Nutr. 2002 Nov;53(6):509-18. doi: 10.1080/09637480220164352. PMID 12590746
- [Background] Heiss C, Kleinbongard P, Dejam A, Perre S, Schroeter H, Sies H, Kelm M. Acute consumption of flavanol-rich cocoa and the reversal of endothelial dysfunction in smokers. J Am Coll Cardiol. 2005 Oct 4;46(7):1276-83. doi: 10.1016/j.jacc.2005.06.055. PMID 16198843
- [Background] Holt RR, Lazarus SA, Sullards MC, Zhu QY, Schramm DD, Hammerstone JF, Fraga CG, Schmitz HH, Keen CL. Procyanidin dimer B2 [epicatechin-(4beta-8)-epicatechin] in human plasma after the consumption of a flavanol-rich cocoa. Am J Clin Nutr. 2002 Oct;76(4):798-804. doi: 10.1093/ajcn/76.4.798. PMID 12324293
- [Background] McKenzie ME, Malinin AI, Bell CR, Dzhanashvili A, Horowitz ED, Oshrine BR, Atar D, Serebruany VL. Aspirin inhibits surface glycoprotein IIb/IIIa, P-selectin, CD63, and CD107a receptor expression on human platelets. Blood Coagul Fibrinolysis. 2003 Apr;14(3):249-53. doi: 10.1097/01.mbc.0000046182.72384.ab. PMID 12695747
- [Background] Tsang C, Auger C, Mullen W, Bornet A, Rouanet JM, Crozier A, Teissedre PL. The absorption, metabolism and excretion of flavan-3-ols and procyanidins following the ingestion of a grape seed extract by rats. Br J Nutr. 2005 Aug;94(2):170-81. doi: 10.1079/bjn20051480. PMID 16115350
- [Background] Tsiara S, Elisaf M, Jagroop IA, Mikhailidis DP. Platelets as predictors of vascular risk: is there a practical index of platelet activity? Clin Appl Thromb Hemost. 2003 Jul;9(3):177-90. doi: 10.1177/107602960300900301. PMID 14507105
- [Background] Williamson G, Manach C. Bioavailability and bioefficacy of polyphenols in humans. II. Review of 93 intervention studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):243S-255S. doi: 10.1093/ajcn/81.1.243S. PMID 15640487